CLINICAL TRIAL: NCT06576193
Title: Empowering Young Parents: Building Health Relationships Study Evaluation of the Safe Dates for Young Parents Intervention
Brief Title: Empowering Young Parents: Building Healthy Relationships Study
Acronym: EYP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TP2AH000082
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Gender-based Violence; Intimate Partner Violence
Keywords: Young Adult Parents; Adolescent Pregnancy; Adolescent Parents; Healthy Relationships

STUDY DESIGN:
Intervention Model Description: Individual AYA will be block-randomized to the SDYP intervention with standard prenatal and post-partum services (intervention condition) or standard services only (control condition) using a 1:1 allocation within each site (stratified randomization) to ensure balanced assignment, using permuted blocks sizes of 4 and 6.
Who Masked: Outcomes Assessor
Masking Description: Field Data Collectors (FDCs) will be masked to the participant group assignments until after the baseline data collection is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe Dates for Young Parents (SDYP) (Experimental): Participants will receive and complete SDYP intervention activities focused on healthy relationships and intimate partner violence (IPV) prevention plus standard services offered at the study site.
  Interventions: Behavioral: Safe Dates for Young Parents (SDYP)
- Standard Services Only (No Intervention): Participants will only receive standard-of-care programming that typically includes services such as one-on-one strength-based case management and comprehensive sex education. The standard services will not address IPV or healthy relationships content that composes the SDYP intervention. Referrals to additional services will be offered to all participants, as needed.

INTERVENTIONS:
Behavioral: Safe Dates for Young Parents (SDYP) — SDYP is a healthy relationship and intimate partner violence (IPV) prevention program, adapted from "Safe Dates (Foshee et al., 1998; Foshee et al., 1996)" designed for teens, that focuses on pregnant or parenting females. The program consists of ten group-based sessions (50 minutes each) led by a trained facilitator which include interactive discussions, analysis of scenarios, games, role-plays, brainstorming, and a poster contest and theatrical play.
  Arms: Safe Dates for Young Parents (SDYP)

SUMMARY:
The goal of this trial is to learn how the Safe Dates for Young Parents (SDYP) intervention affects the sexual and reproductive health behaviors, and quality of, and attitudes surrounding intimate partner relationships in adolescents and young adults (AYA) assigned female sex at birth who are pregnant or parenting.

The main questions it aims to answer are:

* Will the SDYP intervention have any effect on the sexual and reproductive health behaviors during the study period?
* Will the SDYP intervention have any effect on the prevention or reduction of intimate partner violence (IPV)?
* Will the SDYP intervention have any effect on the attitudes and beliefs about healthy relationships?

Researchers will compare the behaviors, attitudes, and beliefs about sexual and reproductive health and relationships of participants assigned to the SDYP intervention group to participants assigned to the control (non-SDYP intervention) group to see if there is any difference or changes in those behaviors, attitudes, and beliefs before-and-after or without the SDYP intervention.

Participants in the SDYP intervention will attend ten (10) 50-minute group sessions that will involve interactive discussions, thinking through life-like scenarios, games, role-plays, brainstorming, and a poster contest and theatrical play.

ELIGIBILITY:
Inclusion Criteria:

Adolescent and Young Adult (AYA) [EYP study participants]

* Aged 14-21 years (inclusive) at Screening.
* Assigned female sex at birth.
* Currently pregnant or parenting their child who lives with them at least part-time.
* Able to speak and read English or Spanish.
* Able and willing to provide verbal informed consent for enrollment in the EYP study.
* Able and willing to provide adequate contact/locator information.
* Able and willing to complete protocol requirements, including completion of three study interviews over one year.

Study Facilitators (process evaluation participants)

* Aged 18 years or older.
* Trained and served as a facilitator of the SDYP intervention.
* Able to speak and read English.
* Able and willing to provide verbal informed consent.

Exclusion Criteria:

* Per participant report at Screening or Enrollment, intends to travel away from their geographic area of residence for a time period that would interfere with study participation, including with intervention participation should the participant be randomized to the SDYP intervention.
* Has any other condition that, in the opinion of the Principal Investigator (PI) or their designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Condomless vaginal or anal sex (Month 12) | Three months, Twelve months
  Participant-reported condom use at recalled instances of vaginal or anal sex over the past 3 months and at 12 months follow-up using a standard, self-administered questionnaire.

SECONDARY OUTCOMES:
Condomless vaginal or anal sex (Month 6) | Three months, Six months
  Participant-reported condom use at recalled instances of vaginal or anal sex over the past 3 months and at 6 months follow-up visit using a standard, self-administered questionnaire.
Sexual and Reproductive Coercion | Month 12
  Participant-reported occurrence of sexual and reproductive coercion with their primary or recent sexual partner at study Month 12 using a 5-point Likert scale questionnaire.
Negotiation of condom use and contraception | Month 6
  Participant-reported ability to successfully negotiate condom and contraceptive-use with their primary or recent sexual partner at study Month 6 using 5- and 4-point Likert scale self-administered questionnaires.
Intimate Partner Violence (IPV) | Month 12
  Participant-reported history, frequency, and severity of IPV (physical and psychological) at study Month 12 using polar (Yes/No), 5- and 4-point Likert scale self-administered questionnaires.
Healthy relationship attitudes, beliefs, and behaviors | Month 6
  Participant-reported attitudes, beliefs, and behaviors about healthy relationships (conflict management skills and emotion regulation) for themselves, their families, or in general at study Month 6 using 5- and 4-point Likert scale self-administered questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Marni Kan, PhD, Study Director — RTI International; Alexandra Minnis, PhD, Principal Investigator — RTI International
Locations (12):
- United States (12):
  - Delaware Adolescent Program, Inc. (DAPI) - Kent County, Camden, Delaware
  - Delaware Adolescent Program, Inc. (DAPI) - Sussex County, Georgetown, Delaware
  - Healthy Generations Program at Children's National Hospital, Washington D.C., District of Columbia
  - GCAPP and Communities In Schools of Albany/Dougherty, Albany, Georgia
  - GCAPP and Covenant House Georgia, Atlanta, Georgia
  - Berrien County Health Department, Benton Harbor, Michigan
  - Eaton Regional Education Service Agency (RESA), Charlotte, Michigan
  - Pathways Academy, Detroit, Michigan
  - Saginaw Intermediate School District, Saginaw, Michigan
  - The Exchange Club, Graham, North Carolina
  - Children & Family Resource Center, Hendersonville, North Carolina
  - Empowering Connections, Partnership for Children & Families, Sanford, North Carolina

IPD SHARING:
Plan to Share IPD: No